CLINICAL TRIAL: NCT06945497
Title: School-based Practices in Arts and Resilience for Kids (SPARK Study)
Brief Title: School-based Practices in Arts and Resilience for Kids
Acronym: SPARK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Chandler Park Academy (Unknown); Jefferson Middle School (Unknown); Lakeview Public Schools (Unknown)
Responsible Party: Principal Investigator, Lana Ruvolo Grasser, Assistant Professor, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 25-02-7541
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Anxiety; Posttraumatic Stress Disorder; Trauma
Keywords: Adversity; Trauma; Stress; Anxiety; Posttraumatic Stress Disorder; Art Therapy; Yoga; Mindfulness; Child and Adolescent
MeSH Terms: conditions — Anxiety Disorders; Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Art Therapy, Yoga/Mindfulness (Experimental): In this arm, participants will first engage in art therapy, then yoga/mindfulness interventions.
  Interventions: Behavioral: Art Therapy; Behavioral: Yoga/Mindfulness
- Yoga/Mindfulness, Art Therapy (Experimental): In this arm, participants will first engage in yoga/mindfulness, then art therapy interventions.
  Interventions: Behavioral: Art Therapy; Behavioral: Yoga/Mindfulness

INTERVENTIONS:
Behavioral: Art Therapy — The art therapy program will include different weekly experientials to explore mindfulness, establish safety, cultivate relaxation, find strength, honor self-identity, and cultivate community. Art media will include markers, colored pencils, fabrics, watercolors, collage, and yarn.
Behavioral: Yoga/Mindfulness — The yoga/mindfulness curriculum will explore consciousness (awareness of self and others), compassion, confidence, courage, and community. Each week, new movement and breathing exercises will be learned.

SUMMARY:
This proposal will implement and test feasibility and efficacy of school-based art therapy and yoga/mindfulness programming to reduce mental health disparities and foster resilience in youth. We will conduct a cross-over randomized trial with n=250 youth (any race/ethnicity or gender, ages 11-14) from two schools: one serving majority Black/African American students and one serving a population-representative ethnoracial demographic with 50% economically disadvantaged students. Baseline data collection will assess experiences of discrimination, negative experiences, positive experiences, and severity of posttraumatic stress, anxiety, depression, somatic symptoms, and resilience. Youth will be randomly assigned to art therapy or yoga/mindfulness for a quarter. Hour-long weekly sessions will occur during elective course times within school to bolster accessibility and generate data to inform future school-based care models for sustainability. Target schools co-developed this design with the research team. At the end of the quarter, participants will engage in post-intervention data collection, including qualitative interviews regarding their experience with the school-based programming. Participants will then cross over to the yoga/mindfulness or art therapy for the subsequent quarter, such that all participants receive both modalities. The methods described above will be repeated, including the assessments. Academic performance will be assessed throughout. We hypothesize that both modalities will be effective in reducing stress, anxiety, and depression related to discrimination, adversity, and trauma that disproportionately impacts racially and ethnically minoritized youth. We anticipate that qualitative feedback will identify points of optimization for programming and inform which students may be most responsive to what intervention(s).

DETAILED DESCRIPTION:
Early life experiences impact development and have lasting effects on health and behavior. Negative childhood experiences (adversity, trauma; e.g., caregiver neglect or maltreatment, community violence, forced migration, discrimination, and harassment, increase the risk for negative mental health outcomes across the lifespan. These negative mental health outcomes include, but are not limited to, posttraumatic stress, anxiety, depression, pain, psychosis, suicidality, and other variation in variation in cognition and emotions. Negative childhood experiences, resultant physical and mental health problems, and associated treatment barriers disproportionately impact racially and ethnically minoritized (non-white) individuals. These disparities are, in part, resultant of historical systemic oppression, exclusion from economic opportunity, lack of representation in healthcare research, and intergenerational trauma exposure. Vulnerability to negative health outcomes may be driven by adversity-driven changes in neural pathways critical for emotion regulation, attention, memory processing, and other cognitive functions. These neural pathways are potentially modifiable with treatment, especially during more flexible developmental windows like childhood and adolescence. Given this, and that most psychiatric disorders onset in childhood or adolescence, the school age is the best time to intervene to mitigate future physical, mental, educational, and socioeconomic consequences of negative childhood experiences.

Barriers to accessing mental health care include lack of transportation, financial concerns, negative expectations surrounding seeking mental health services, medical mistrust rooted in historical injustice and trauma, and stigma. Therefore, there is a great need to facilitate healthy biopsychosocial development of youth by fostering resilience. Resilience, in part, is the ability to cope when faced with adversity. Cultivating resilience can protect against the negative impacts of childhood adversity. Fostering resilience can be achieved by teaching youth how to manage stress, regulate emotions and reactions, and resolve interpersonal disputes. One strategy to accomplish this at scale is by implementing school-based programs that support social-emotional learning. Expanding access to care and improving opportunities for youth via school-based mental health services can reduce disparities. Current gold-standard psychotherapy (e.g., cognitive behavioral therapy) and medication (e.g., serotonin-selective reuptake inhibitors) treat symptoms rather than cultivate resilience and are limited by availability, cost, accessibility, and adherence, especially for children and from individuals from disadvantaged backgrounds. Additionally, up to 50% of patients do not adequately respond to these treatments. These care models center around reactive, rather than proactive, care models based on research from predominantly white, highly educated, high socioeconomic status individuals. There is a need for a more diverse approach to methods of improving mental health with broader access for the general population and prevention/early interventions. Therefore, identifying accessible and cost-effective ways to reduce psychopathology and cultivate resilience in youth is a high priority to curb the myriad negative physical health, socioemotional, and economic sequelae.

To address the barriers to traditional forms of therapeutic care in youth, school-based art therapy and yoga/mindfulness pose as well-suited options. Art therapy, yoga, and mindfulness are interventions that target emotion (dys)regulation by integrating experientials that probe creativity, flexibility, and adaptability to better develop cognitive flexibility. Therapies that enhance emotion regulation and target underlying neural circuits may confer greater ability to dampen reactivity to stress and negative experiences. By offering these interventions in a group setting, school-based art therapy and yoga/mindfulness also has the opportunity to cultivate social support and peer interactions-fostering protective factors that have been found to reduce risk for mental illness in children and adolescents in a cost-effective and accessible manner. Offering such interventions at the group level may not only benefit those experiencing significant mental distress, but may also benefit those who are not experiencing such symptoms, as they will still reap the long-term benefits of building stress-relaxation and emotion regulation coping skills. Art therapy and yoga/mindfulness have all shown promise for reducing trauma, stress, anger, depression, obsessive compulsiveness, and anxiety.

One strategy to overcome mental healthcare barriers (e.g., transportation, finances, and stigma) and foster resilience in youth is to implement school-based programs that support social and emotional development. Art therapy and yoga/mindfulness have similar therapeutic goals to help children feel a sense of control and structure and reduce stress. Art therapy and yoga/mindfulness help children with self-regulation, resilience and promote well-being through increased awareness, healthy behaviors, and stress management in a cost-effective and accessible manner.The significant impact of these interventions will encourage a greater diversity of patients, physicians, and communities to participate in and support use of arts and mindfulness interventions as a main mode of cost-effective and accessible treatment.

The present proposal is directly responsive to Senate Resolution 769 from the 118th Congress to "support student well-being through evidence-based prevention strategies" give the gross "lack [of] adequate services and support when dealing with mental health challenges and crises." School and community settings offer viable venues for broad-scale implementation of interventions. Art therapy and yoga/mindfulness may be favorable for youth implemented in schools and community settings for a) augmenting healthcare services youth may receive, b) providing an accessible and affordable option for youth untreated due to lack of access to care, cost, or stigmatization, and c) instill coping skills and relaxation techniques in youth who have experienced adversity and discrimination.

Vulnerability to negative health outcomes may be driven by adversity-driven changes in neural pathways critical for emotion regulation, attention, memory processing, and other cognitive functions. These neural pathways are potentially modifiable with treatment, especially during more flexible developmental windows like childhood and adolescence. Given this, and that most psychiatric disorders onset in childhood or adolescence, the school age is the best time to intervene to mitigate future physical, mental, educational, and socioeconomic consequences of negative childhood experiences.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 11-14 years, inclusive.
2. Any gender identity or sex assigned at birth.
3. English-speaking, given that study interventions and assessments will be in English.
4. Ability to provide written informed assent or oral assent.
5. Caregiver ability to provide informed consent and ability to assist in completing study.
6. Student enrolled in collaborating school.

Note: here, we define 'caregiver' as the participant's parent and/or legal guardian.

Exclusion Criteria:

1. Current or past bipolar I/II disorder
2. Current or past psychotic disorder
3. Autism spectrum disorders or any other severe developmental disorder

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Anxiety | One year
  We will measure severity of self-reported anxiety symptoms before, during, and after interventions, up to 3 months post interventions, for a total duration of one year. To measure severity of self-reported anxiety symptoms, we will use the Screen for Child Anxiety-Related Emotional Disorders, a valid and reliable measure for children and adolescents ages 7-17. The SCARED captures symptoms related to panic disorder / somatic symptoms, generalized anxiety disorder, separation anxiety, social anxiety, and school avoidance.

SECONDARY OUTCOMES:
Posttraumatic Stress | One year
  We will measure severity of self-reported post traumatic stress symptoms in youth who endorse at least one traumatic exposure. To measure traumatic exposures and PTSD symptoms, we will use the UCLA PTSD Reaction Index. The UCLA PTSD RI is a valid and reliable measure developed for children and adolescents ages 7-17. The first component of the measures captures the index trauma (Criterion A), and the second component assesses the core symptoms of PTSD - reexperiencing / intrusive symptoms (Criterion B), avoidance (Criterion C), negative changes in cognitions and mood (Criterion D), arousal (Criterion E), and dissociative symptoms (Dissociative Subtype). We will measure symptoms before, during, and after the intervention, up to three months post interventions, for a total duration of one year.
Depression | One year
  We will measure self-reported severity of depression. To measure self-reported severity of depression, we will use the Mood and Feelings Questionnaire. The Mood and Feelings Questionnaire is a valid and reliable measure for assessing symptoms related to depression in children and adolescents. We will measure symptoms before, during, and after the intervention, up to three months post interventions, for a total duration of one year.
Resilience | One year
  We will measure self-reports of resilience using the Brief Resilience Scale. We will measure resilience before, during, and after the intervention, up to three months post interventions, for a total duration of one year.

CONTACTS AND LOCATIONS:
Overall Officials: Lana R Grasser, Ph.D., Principal Investigator — Wayne State University
Locations (2):
- United States (2):
  - Chandler Park Academy Middle School, Harper Woods, Michigan
  - Jefferson Middle School, Saint Clair Shores, Michigan

IPD SHARING:
Plan to Share IPD: Yes
De-identified data that does not include any personal identifying information (e.g., date of birth, social security number, contact information, names, etc.) will be shared. This includes, but is not limited to, non-PII demographic information, reports of positive and negative (e.g., discrimination, adversity, trauma) experiences, severity of self-reported anxiety, depression, and post traumatic stress disorder, and resilience. Item-level as well as scored data will be shared according to published guidelines.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We will share IPD and supporting information within three years of the end date of data collection. Data will be shared indefinitely (no end date), unless individual participants choose to withdraw their data from data sharing.
Access Criteria: IPD and supporting information will be publicly accessible via GitHub, an online website that is free/open source.
URL: https://github.com

REFERENCES:
- [Background] Grasser LR, Marusak H. Strong Mind, Strong Body: The Promise of Mind-Body Interventions to Address Growing Mental Health Needs Among Youth. Mental Health Sci. 2023 Jun;1(2):58-66. doi: 10.1002/mhs2.16. Epub 2023 Mar 22. PMID 37810896
- [Background] Lesté A, Rust J. Effects of dance on anxiety. American Journal of Dance Therapy. 1990/03/01 1990;12(1):19-25. doi:10.1007/BF00844312
- [Background] Lee H-J, Jang S-H, Lee S-Y, Hwang K-S. Effectiveness of dance/movement therapy on affect and psychotic symptoms in patients with schizophrenia. The Arts in Psychotherapy. 2015/09/01/ 2015;45:64-68. doi:https://doi.org/10.1016/j.aip.2015.07.003
- [Background] Grasser LR, Al-Saghir H, Wanna C, Spinei J, Javanbakht A. Moving Through the Trauma: Dance/Movement Therapy as a Somatic-Based Intervention for Addressing Trauma and Stress Among Syrian Refugee Children. J Am Acad Child Adolesc Psychiatry. 2019 Nov;58(11):1124-1126. doi: 10.1016/j.jaac.2019.07.007. Epub 2019 Jul 23. PMID 31348987
- [Background] Feen-Calligan H, Ruvolo Grasser L, Debryn J, et al. Art therapy with Syrian refugee youth in the United States: An intervention study. The Arts in Psychotherapy. 2020/07/01/ 2020;69:101665. doi:https://doi.org/10.1016/j.aip.2020.101665
- [Background] Feder A, Fred-Torres S, Southwick SM, Charney DS. The Biology of Human Resilience: Opportunities for Enhancing Resilience Across the Life Span. Biol Psychiatry. 2019 Sep 15;86(6):443-453. doi: 10.1016/j.biopsych.2019.07.012. Epub 2019 Jul 24. PMID 31466561
- [Background] Brown EC, Graham JW, Hawkins JD, Arthur MW, Baldwin MM, Oesterle S, Briney JS, Catalano RF, Abbott RD. Design and analysis of the Community Youth Development Study longitudinal cohort sample. Eval Rev. 2009 Aug;33(4):311-34. doi: 10.1177/0193841X09337356. Epub 2009 Jun 9. PMID 19509119
- [Background] Lerner RM, Lerner JV, Almerigi JB, et al. Positive youth development, participation in community youth development programs, and community contributions of fifth grade adolescents: findings from the First Wave of the 4-H Study of Positive Youth Development. The Journal of Early Adolescence. 2005;25:17-71.
- [Background] Minton SC, Faber R. Thinking with the Dancing Brain: Embodying Neuroscience. Rowman & Littlefield; 2016.
- [Background] Bailey JM, Bartlem KM, Wiggers JH, Wye PM, Stockings EAL, Hodder RK, Metse AP, Regan TW, Clancy R, Dray JA, Tremain DL, Bradley T, Bowman JA. Systematic review and meta-analysis of the provision of preventive care for modifiable chronic disease risk behaviours by mental health services. Prev Med Rep. 2019 Aug 14;16:100969. doi: 10.1016/j.pmedr.2019.100969. eCollection 2019 Dec. PMID 31497500
- [Background] Henrich J, Heine SJ, Norenzayan A. Most people are not WEIRD. Nature. 2010 Jul 1;466(7302):29. doi: 10.1038/466029a. No abstract available. PMID 20595995
- [Background] Alegría M, Green JG, McLaughlin KA, Loder S. Disparities in child and adolescent mental health and mental health services in the US. New York, NY: William T Grant Foundation. 2015:26.
- [Background] Hampton-Anderson JN, Carter S, Fani N, Gillespie CF, Henry TL, Holmes E, Lamis DA, LoParo D, Maples-Keller JL, Powers A, Sonu S, Kaslow NJ. Adverse childhood experiences in African Americans: Framework, practice, and policy. Am Psychol. 2021 Feb-Mar;76(2):314-325. doi: 10.1037/amp0000767. PMID 33734797
- [Background] Slopen N, Shonkoff JP, Albert MA, Yoshikawa H, Jacobs A, Stoltz R, Williams DR. Racial Disparities in Child Adversity in the U.S.: Interactions With Family Immigration History and Income. Am J Prev Med. 2016 Jan;50(1):47-56. doi: 10.1016/j.amepre.2015.06.013. Epub 2015 Sep 2. PMID 26342634
- [Background] Bremner JD, Ortego RA, Campanella C, Nye JA, Davis LL, Fani N, Vaccarino V. Neural correlates of PTSD in women with childhood sexual abuse with and without PTSD and response to paroxetine treatment: A placebo-controlled, double-blind trial. J Affect Disord Rep. 2023 Dec;14:100615. doi: 10.1016/j.jadr.2023.100615. Epub 2023 Jun 24. PMID 38088987
- [Background] Henrich J, Heine SJ, Norenzayan A. The weirdest people in the world? Behav Brain Sci. 2010 Jun;33(2-3):61-83; discussion 83-135. doi: 10.1017/S0140525X0999152X. Epub 2010 Jun 15. PMID 20550733
- [Background] Waldman SA, Terzic A. Health Care Evolves From Reactive to Proactive. Clin Pharmacol Ther. 2019 Jan;105(1):10-13. doi: 10.1002/cpt.1295. PMID 30597564
- [Background] Grasser LR, Jovanovic T. Neural Impacts of Stigma, Racism, and Discrimination. Biol Psychiatry Cogn Neurosci Neuroimaging. 2022 Dec;7(12):1225-1234. doi: 10.1016/j.bpsc.2022.06.012. Epub 2022 Jul 8. PMID 35811064
- [Background] Grasser LR, Jovanovic T. Safety learning during development: Implications for development of psychopathology. Behav Brain Res. 2021 Jun 25;408:113297. doi: 10.1016/j.bbr.2021.113297. Epub 2021 Apr 18. PMID 33862062
- [Background] Cross D, Fani N, Powers A, Bradley B. Neurobiological Development in the Context of Childhood Trauma. Clin Psychol (New York). 2017 Jun;24(2):111-124. doi: 10.1111/cpsp.12198. Epub 2017 May 20. PMID 30906116
- [Background] Fani N, Stenson AF, van Rooij SJH, La Barrie DL, Jovanovic T. White matter microstructure in trauma-exposed children: Associations with pubertal stage. Dev Sci. 2021 Nov;24(6):e13120. doi: 10.1111/desc.13120. Epub 2021 May 13. PMID 33983665
- [Background] Webb EK, Harnett NG. The biological embedding of structural inequities: new insight from neuroscience. Neuropsychopharmacology. 2024 Jan;49(1):337-338. doi: 10.1038/s41386-023-01655-8. No abstract available. PMID 37463977
- [Background] Fani N, White D, Marshall-Lee E, Hampton-Anderson J. Antiracist Practice in Psychiatry: Principles and Recommendations. Focus (Am Psychiatr Publ). 2022 Jul;20(3):270-276. doi: 10.1176/appi.focus.20220045. Epub 2022 Jul 1. PMID 37205017
- [Background] Powers A, Fani N, Cross D, Ressler KJ, Bradley B. Childhood trauma, PTSD, and psychosis: Findings from a highly traumatized, minority sample. Child Abuse Negl. 2016 Aug;58:111-8. doi: 10.1016/j.chiabu.2016.06.015. Epub 2016 Jun 29. PMID 27371800
- [Background] Ginty AT, Kraynak TE, Fisher JP, Gianaros PJ. Cardiovascular and autonomic reactivity to psychological stress: Neurophysiological substrates and links to cardiovascular disease. Auton Neurosci. 2017 Nov;207:2-9. doi: 10.1016/j.autneu.2017.03.003. Epub 2017 Mar 16. PMID 28391987
- [Background] Nicolaides NC, Kyratzi E, Lamprokostopoulou A, Chrousos GP, Charmandari E. Stress, the stress system and the role of glucocorticoids. Neuroimmunomodulation. 2015;22(1-2):6-19. doi: 10.1159/000362736. Epub 2014 Sep 12. PMID 25227402
- [Background] Akil H. Stressed and depressed. Nat Med. 2005 Feb;11(2):116-8. doi: 10.1038/nm0205-116. No abstract available. PMID 15692589
- [Background] Ainamani HE, Weierstall-Pust R, Bahati R, Otwine A, Tumwesigire S, Rukundo GZ. Post-traumatic stress disorder, depression and the associated factors among children and adolescents with a history of maltreatment in Uganda. Eur J Psychotraumatol. 2022 Jan 10;13(1):2007730. doi: 10.1080/20008198.2021.2007730. eCollection 2022. PMID 35028113
- [Background] Gazendam FJ, Krypotos AM, Kamphuis JH, van der Leij AR, Huizenga HMH, Eigenhuis A, Kindt M. From adaptive to maladaptive fear: Heterogeneity in threat and safety learning across response systems in a representative sample. Int J Psychophysiol. 2020 Dec;158:271-287. doi: 10.1016/j.ijpsycho.2020.09.017. Epub 2020 Oct 17. PMID 33080297